CLINICAL TRIAL: NCT04618783
Title: Cross-neutralization Capacity of Immune Serum From Different Dosage of Sabin Inactivated Poliovirus Vaccine Immunization Against Multiple Individual Wild and Vaccine-derived Polioviruses, Supplementary Study of a Phase 2 Clinical Trial.
Brief Title: Cross-neutralization Capacity of Immune Serum From Different Dosage of Sabin Inactivated Poliovirus Vaccine Immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-sIPV-1001-1
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dosage experimental group (Experimental): Three doses of low-dosage investigational sIPV, vaccinated within one-month interval between doses
  Interventions: Biological: Three doses of low-dosage investigational sIPV, vaccinated within one-month interval between doses
- Medium-dosage experimental group (Experimental): Three doses of medium-dosage investigational sIPV, vaccinated within one-month interval between doses
  Interventions: Biological: Three doses of medium-dosage investigational sIPV, vaccinated within one-month interval between doses
- High-dosage experimental group (Experimental): Three doses of high-dosage investigational sIPV, vaccinated within one-month interval between doses
  Interventions: Biological: Three doses of high-dosage investigational sIPV, vaccinated within one-month interval between doses
- Control wIPV group (Active Comparator): Three doses of control wIPV, vaccinated within one-month interval between doses
  Interventions: Biological: Three doses of control wIPV, vaccinated within one-month interval between doses
- Control sIPV group (Active Comparator): Three doses of control sIPV, vaccinated within one-month interval between doses
  Interventions: Biological: Three doses of control sIPV, vaccinated within one-month interval between doses

INTERVENTIONS:
Biological: Three doses of low-dosage investigational sIPV, vaccinated within one-month interval between doses — Antigen content: 7.5, 22.5, and 22.5 D-antigen unite for type 1, 2, and 3 in 0.5 ml diluent per dose
  Arms: Low-dosage experimental group
Biological: Three doses of medium-dosage investigational sIPV, vaccinated within one-month interval between doses — Antigen content: 15, 45, and 45 D-antigen unite for type 1, 2, and 3 in 0.5 ml diluent per dose
  Arms: Medium-dosage experimental group
Biological: Three doses of high-dosage investigational sIPV, vaccinated within one-month interval between doses — Antigen content: 22.5, 67.5, and 67.5 D-antigen unite for type 1, 2, and 3 in 0.5 ml diluent per dose
  Arms: High-dosage experimental group
Biological: Three doses of control wIPV, vaccinated within one-month interval between doses — Antigen content: 40, 8, and 32 D-antigen unite for type 1, 2, and 3 in 0.5 ml diluent per dose
  Arms: Control wIPV group
Biological: Three doses of control sIPV, vaccinated within one-month interval between doses — Antigen content: 30, 32, and 45 D-antigen unite for type 1, 2, and 3 in 0.5 ml diluent per dose
  Arms: Control sIPV group

SUMMARY:
This study is a supplementary study of an already finished randomised, double-blinded, and placebo controlled phase 2 clinical trial of an Sabin strain inactivated poliovirus vaccine (sIPV) manufactured by Sinovac Biotech Ltd., Beijing China. The purpose of this study is to evaluate the cross-neutralization capacity of the serum immuned by the investigational sIPV against 10 individual virus strains.

DETAILED DESCRIPTION:
This study is a open-labelled study conducted based on an already finished phase 2 study of the investigational sIPV in 600 healthy infants aged 2-months old. The purpose of this study is to evaluate the cross-neutralization capacity of the serum immuned by the investigational sIPV against 10 individual virus strains. Paired pre-immune and post-immune serum from 250 participants of the phase 2 trial, with 50 in each group including the low-, medium- and high- dosage group, control wild poliovirus vaccine (wIPV) group and control sIPV group, was selected and sent to China Center for Disease Control and Prevention (CDC) for the cross-neutralization assay to determine the neutralizing antibody titer against 10 individual virus strains including Sabin strains (type 1, 2, and 3), Salk strains (Mahoney, MEF-1, and Saukett), cVDPV (type 1, 2, and 3) and Xinjiang wild strain of type 1(Xinjiang wIPV1).

All the subjects in this study had been vaccinated at the schedule of month 0,1, and 2 in the phase 2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the already finished phase 2 clinical trial;
* Subjects who received the three-doses full schedule vaccination required in the phase 2 tril and can provide the backup paired pre-immune and post-immune serum collected in the phase trial;
* Provide written informed consent.

Exclusion Criteria:

* None.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Immunity index of seroconversion rate | One month after three doses of vaccination
  The seroconversion rates of neutralizing antibody against 10 individual virus strains (Sabin 1, Sabin2， Sabin 3, Mahoney 1, MEF-1, Saukett, cVDPV1, cVDPV2, cVDPV3, and Xinjiang wIPV1)

SECONDARY OUTCOMES:
Immunity index of geometric mean titer (GMT) | One month after three doses of vaccination
  The GMT of neutralizing antibody against 10 individual virus strains (Sabin 1, Sabin2， Sabin 3, Mahoney 1, MEF-1, Saukett, cVDPV1, cVDPV2, cVDPV3, and Xinjiang wIPV1)
Immunity index of geometric mean ratio (GMR) | One month after three doses of vaccination
  The GMR of neutralizing antibody against 10 individual virus strains (Sabin 1, Sabin2， Sabin 3, Mahoney 1, MEF-1, Saukett, cVDPV1, cVDPV2, cVDPV3, and Xinjiang wIPV1)
Immunity index of seropositivity rate | One month after three doses of vaccination
  The seropositivity rate of neutralizing antibody against 10 individual virus strains (Sabin 1, Sabin2， Sabin 3, Mahoney 1, MEF-1, Saukett, cVDPV1, cVDPV2, cVDPV3, and Xinjiang wIPV1)

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Pizhou Center for Disease Control and Prevention, Pizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No